CLINICAL TRIAL: NCT05072860
Title: The Adjunctive Role of Temporary Uterine Packing Combined With Topical Tranexamic Acid for the Prevention of Postpartum Hemorrhage in Hypertensive Women Undergoing Elective Cesarean Section: A Randomized Controlled Trial
Brief Title: Topical Tranexamic Acid for the Prevention of Postpartum Hemorrhage in Women Undergoing Elective Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/542/7/21
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: a double-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a double-blinded randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical tranexamic acid (Experimental): temporary uterine packing with gauze of the dimensions soaked with 2 gm tranexamic diluted in 60ml saline acid or placebo
  Interventions: Drug: Topical tranexamic acid
- normal saline (Placebo Comparator): temporary uterine packing with gauze of the dimensions soaked with 2 gm placebo to tranexamic diluted in 60ml saline acid
  Interventions: Other: : normal saline

INTERVENTIONS:
Drug: Topical tranexamic acid — temporary uterine packing with gauze of the dimensions soaked with 2 gm tranexamic diluted in 60ml saline acid
  Other Names: experimental
  Arms: Topical tranexamic acid
Other: : normal saline — temporary uterine packing with gauze of the dimensions soaked with placebo to 2 gm tranexamic diluted in 60ml saline acid
  Other Names: Placebo Comparator
  Arms: normal saline

SUMMARY:
In hypertensive women having an elective cesarean section, the effectiveness and safety of temporary uterine packing coupled with topical tranexamic acid as an adjuvant for decreasing blood loss during delivery were compared to placebo.

DETAILED DESCRIPTION:
patients were allocated to one of two groups after induction of anesthesia. they received temporary uterine packing with gauze of the dimensions soaked with 2 gm tranexamic diluted in 60ml saline acid or placebo

ELIGIBILITY:
Inclusion Criteria:

* hypertensive women undergoing elective cesarean section

Exclusion Criteria:

* Patients with cardiac, hepatic, renal, or thromboembolic disease. ,
* patients with the high possibility of the morbid adherent placenta,
* known coagulopathy and
* those presented with severe antepartum hemorrhage
* refuse to participate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — hypertensive women undergoing elective cesarean section
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | 30 minutes
  measures the intraoperative blood loss by direct and gravimetric methods

SECONDARY OUTCOMES:
need of blood transfusion | 12 hours
  number of unites of blood transfusion
need of uterotonic | 24 hours
  misoprostol, oxytocin etc
change in hemoglobin | 24 hours
  change in hemoglobin

IPD SHARING:
Plan to Share IPD: No